CLINICAL TRIAL: NCT01092962
Title: Cyclophosphamide Versus Mycophenolate Mofetil for Children With Steroid-dependent Idiopathic Nephrotic Syndrome : a Multicenter Randomized Controlled Trial
Brief Title: Cyclophosphamide Versus Mycophenolate Mofetil for the Treatment of Steroid-dependent Nephrotic Syndrome in Children
Acronym: NEPHROMYCY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P071221
Record Dates: First submitted 2010-02-26; First posted 2010-03-25 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2013-08

CONDITIONS: Idiopathic Nephrotic Syndrome
Keywords: Children; Mycophenolate mofetil; Cyclophosphamide; Idiopathic nephrotic steroid sensitive syndrome
MeSH Terms: conditions — Nephrosis, Lipoid | interventions — Cyclophosphamide; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycophenolate mofetil (Experimental): Mycophenolate mofetil
  Interventions: Drug: Mycophenolate mofetil
- Cyclophosphamide (Active Comparator): Cumulative dose of 148mg/kg of cyclophosphamide in 84 days (2mg/kg/day during 12 weeks)
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — 2mg/kg/day during 12 weeks (cumulative dose 148mg/kg)
  Other Names: Endoxan (BAXTER)
  Arms: Cyclophosphamide
Drug: Mycophenolate mofetil — 1200mg/m²/jour in two divided doses during 18 months
  Other Names: Cellcept (Roche)
  Arms: Mycophenolate mofetil

SUMMARY:
Idiopathic nephrotic syndrome is steroid-sensitive in more than 90% of cases in children. However 60% of cases are steroid dependent and required treatment with immunosuppressive agent. Cyclophosphamide and ciclosporin are used for long time to reduce steroid dependency, but duration of these treatments should be restricted because of gonadotoxicity for cyclophosphamide and nephrotoxicity for ciclosporin.

Mycophenolate mofetil appears as an alternative treatment without gonadotoxicity and nephrotoxicity. However, contrary to cyclophosphamide, mycophenolate mofetil does not seem to have a residual action so that treatment must be maintained during months or years.

The aim of the study is to compare efficacy of cyclophosphamide and mycophenolate mofetil in steroid dependent nephrotic syndrome in children.

DETAILED DESCRIPTION:
Aim of the study: Comparison of efficacy of cyclophosphamide 148mg/kg in 12 weeks and mycophenolate mofetil 1200mg/m² during 18 months, in children with steroid dependent nephrotic syndrome.

The 70 patients will be recruited in the 26 centres of paediatric nephrology in France, included and randomized at the time of a relapse. They will receive the same steroid treatment in the 2 arms.

The primary point will be occurrence of a relapse during the 24 months of follow-up. Detection of relapse will be done by using dipsticks and confirm by biological dosages (albuminemia and proteinuria/CREATININURIA ratio). Clinical and biological check up will be done every 3 months during all the study.

ELIGIBILITY:
Inclusion Criteria:

* children 2 to 16 years old
* steroid dependency ≥30mg/m² eod
* or steroid dependency ≥15mg/m² eod and occurrence of : at least 2 relapses in 1 year, adverse event of steroid therapy (height rate ≤-1SD, obesity, other complication) or severe complication of nephrotic syndrome (thrombosis, collapse, severe infection,…)
* inform consent

Exclusion Criteria:

* steroid resistant nephrotic syndrome
* prior treatment with cyclophosphamide, mycophenolate mofetil or cyclosporine
* absence of contraception in pubescent girls
* allergy to cyclophosphamide or mycophenolate mofetil
* malignant disease
* treatment with other immunosuppressant treatment or with non-steroid anti-inflammatory or anti proteinuric medication (enzyme converse antagonist and angiotensin II receptor antagonist)
* absence of inform consent
* participation to other therapeutic trial

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2010-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Relapse of nephrotic syndrome (defined by occurrence of proteinuria ≥ 0,25 g/mmol of CREATININURIA (or ≥ 2g/g) with hypoalbuminemia ≤ 30g/L AND/OR dipsticks >2+ during 3 days and proteinuria/CREATININURIA ratio ≥ 0,25 g/mmol) during 2 years. | Months 1, 3, 6, 9, 12, 15, 18, 21, 24

SECONDARY OUTCOMES:
In case of relapse, steroid threshold dose to maintain a remission compare to those before inclusion in the study | Months 1, 3, 6, 9, 12, 15, 18, 21, 24
Cumulative steroid dose received during the years before and under treatment | Months 1, 3, 6, 9, 12, 15, 18, 21, 24
Comparison of growth data, during the year before and under treatment | Months 1, 3, 6, 9, 12, 15, 18, 21, 24
Pharmacokinetics measurement of MPA and relation with efficacy in case of treatment with MMF | One month after beginning MMF

CONTACTS AND LOCATIONS:
Overall Officials: Véronique BAUDOUIN, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, AP-HP, Paris, Paris, France

REFERENCES:
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526